CLINICAL TRIAL: NCT05310994
Title: Efficacy Evaluation of Wasabi (Wasabia Japonica) Leaf Extract on Skin
Brief Title: Efficacy Evaluation of Wasabi Leaf Extract on Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CMUH111-REC3-028
Record Dates: First submitted 2022-03-28; First posted 2022-04-05 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Skin Condition
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo drink (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo drink
- Wasabi Leaf Extract Drink (Experimental)
  Interventions: Dietary Supplement: Wasabi Leaf Extract Drink

INTERVENTIONS:
Dietary Supplement: Placebo drink — consume 1 bottle per day
  Arms: Placebo drink
Dietary Supplement: Wasabi Leaf Extract Drink — consume 1 bottle per day
  Other Names: Wasabi (Wasabia japonica) leaf extract drink
  Arms: Wasabi Leaf Extract Drink

SUMMARY:
To assess the efficacy of Wasabi Leaf Extract on skin

ELIGIBILITY:
Inclusion Criteria:

* 20 to 65-year-old males or females
* People with dull skin, pigmentation spots or acne-prone, acne scars
* Acne severity assessment- Investigator's Global Assessment Scale (IGA) ≥ 2

Exclusion Criteria:

* Received medical cosmetic treatment (including cosmetic skin care, laser, fruit acid peeling, injection or plastic surgery, etc.) currently or within one month before the trial
* Outdoor workers (exposed to the sun more than 5 hours a day)
* People who are breastfeeding, pregnant or planning to become pregnant during the test (self-report)
* People with heart, liver, kidney, endocrine and other major organic diseases (self-reported)
* People who have undergone major surgery (according to medical history)
* People who take drugs for a long time
* People with mental illness
* Students who are currently taking courses taught by the principal investigator of this trial

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
The change of skin melanin index | Change from Baseline skin melanin index at 8 weeks
  Mexameter® MX18 was utilized to measure skin melanin index. Units: arbitrary Mexameter® units (0-999)
The change of skin erythema index | Change from Baseline skin erythema index at 8 weeks
  Mexameter® MX18 was utilized to measure skin erythema index. Units: arbitrary Mexameter® units (0-999)
The change of skin sebum content | Change from Baseline skin sebum content at 8 weeks
  Sebumeter® SM815 was utilized to measure skin sebum content. Units: Sebumeter® units from 0-350
The change of transepidermal water loss | Change from Baseline TEWL at 8 weeks
  Tewameter® TM300 was utilized to measure transepidermal water loss (TEWL). Units: TEWL-values lower than 70 g/hm²
The change of L* (lightness) values | Change from Baseline L* value at 8 weeks
  Spectrophotometer SCM-108 was utilized to measure skin L* value. Units: arbitrary units
The change of a* (redness) values | Change from Baseline a* value at 8 weeks
  Spectrophotometer SCM-108 was utilized to measure skin a* value. Units: arbitrary units
The change of visible spots | Change from Baseline visible spots at 8 weeks
  VISIA Complexion Analysis System was utilized to measure skin spots. Units: arbitrary units
The change of skin red area | Change from Baseline skin red area at 8 weeks
  VISIA Complexion Analysis System was utilized to measure skin red area. Units: arbitrary units
The change of total antioxidant capacity of blood | Change from Baseline total antioxidant capacity at 8 weeks
  Venous blood was sampled to measure total antioxidant capacity
The change of Interleukin-6 of blood | Change from Baseline IL-6 at 8 weeks
  Venous blood was sampled to measure IL-6
The change of Interleukin-8 of blood | Change from Baseline IL-8 at 8 weeks
  Venous blood was sampled to measure IL-8
The change of Insulin-Like Growth Factor-1 of blood | Change from Baseline IGF-1 at 8 weeks
  Venous blood was sampled to measure IGF-1

SECONDARY OUTCOMES:
The change of skin hydration | Change from Baseline skin hydration at 8 weeks
  Corneometer® CM825 was utilized to measure skin hydration. Units: arbitrary
The change of UV spots | Change from Baseline UV spots at 8 weeks
  VISIA Complexion Analysis System was utilized to measure UV spots. Units: arbitrary units
The change of brown spots | Change from Baseline brown spots at 8 weeks
  VISIA Complexion Analysis System was utilized to measure brown spots. Units: arbitrary units
The change of Advanced glycation end products of blood | Change from Baseline AGEs at 8 weeks
  Venous blood was sampled to measure AGEs
The change of liver function biomarkers (AST, ALT) of blood | Change from Baseline liver function biomarkers at 8 weeks
  Venous blood was sampled to measure liver function biomarkers
The change of renal function biomarkers (creatinine, BUN) of blood | Change from Baseline renal function biomarkers at 8 weeks
  Venous blood was sampled to measure renal function biomarkers
The change of fasting blood glugose level | Change from Baseline fasting blood glugose level at 8 weeks
  Venous blood was sampled to measure fasting blood glugose level
The change of blood lipid profile | Change from Baseline blood lipid profile at 8 weeks
  Venous blood was sampled to measure blood lipid profile (total cholesterol, HDL-C, LDL-C, triglyceride)

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu-Mei Chiang, Prof., Principal Investigator — China Medical University, China; Po-Yuan Wu, Dr., Study Director — China Medical University Hospital
Locations (1):
- China Medical University, Taichung, Taiwan